CLINICAL TRIAL: NCT04122534
Title: Somatic Mindfulness Training for a Healthy Workforce: Student Pilot Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Kelly Knight, Associate Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1111
Record Dates: First submitted 2019-09-28; First posted 2019-10-10 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Occupational-based Secondary Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Treatment groups receives the intervention training.
  Interventions: Behavioral: Somatic Mindfulness Training

INTERVENTIONS:
Behavioral: Somatic Mindfulness Training — Educational and experiential training to reduce occupational-based secondary trauma.

SUMMARY:
This pilot study evaluates a somatic mindfulness training. Reductions in mental and physical health correlates of secondary trauma are assessed using a pretest-posttest design.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be either employed or volunteering as a victim service provider, or enrolled at Montana State University as an undergraduate student.

Exclusion Criteria:

* Participant is under age 18.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 48
Completed | 44
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.67 (2.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 41
  More than one race | 4
  Unknown or Not Reported | 1
Secondary Traumatic Stress Scale [Mean (Standard Deviation); unit: units on a scale] — Measures occupational-based secondary traumatic stress using a total scale range of 17(min) to 85 (max). Scores above 37 indicate moderate or higher secondary traumatic stress. Population: Missing data.
  units on a scale
    number analyzed (Participants) | 35
    (all) | 35.71 (10.51)
Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Measures symptoms of post-traumatic stress disorder using a total scale range of 0 (min) to 80 (max), with a score of 33 or higher indicating that participants maybe suffering from Post Traumatic Stress Disorder.
  units on a scale | 31.42 (15.86)

OUTCOME MEASURES:

1. Primary Outcome: Secondary Traumatic Stress Scale
Description: Measures occupational-based secondary traumatic stress using a total scale range of 17(min) to 85 (max). Scores above 37 indicate moderate or higher secondary traumatic stress.
Time Frame: This outcome measure will be assessed at week 15.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 26
units on a scale | 35.23 (13.02)

2. Secondary Outcome: Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5)
Description: Measures symptoms of post-traumatic stress disorder using a total scale range of 0 (min) to 80 (max), with a score of 33 or higher indicating that participants maybe suffering from Post Traumatic Stress Disorder.
Time Frame: This outcome measure will be assessed at week 15.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 43
units on a scale | 28.47 (15.35)

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

LIMITATIONS AND CAVEATS:
Outcome measures collected during COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04122534/Prot_SAP_ICF_000.pdf